CLINICAL TRIAL: NCT01071876
Title: BF2.649 in Patients With Obstructive Sleep Apnea Syndrome (OSA) and Treated by Nasal Continuous Positive Airway Pressure (nCPAP), But Still Complaining of Excessive Daytime Sleepiness (EDS)
Brief Title: BF2.649 in Patients With OSA and Treated by CPAP But Still Complaining of EDS
Acronym: HAROSA1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P09-08 / BF2.649; 2009-017248-14 (EudraCT Number)
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Obstructive Sleep Apnea; Excessive Daytime Sleepiness
Keywords: Sleep disorder; obstructive sleep apnea; excessive daytime sleepiness; patients with OSA treated by CPAP presenting EDS
MeSH Terms: conditions — Sleep Apnea, Obstructive; Disorders of Excessive Somnolence; Sleep Wake Disorders | interventions — pitolisant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BF2.649 (Experimental): BF2.649 capsules dosed at 5mg, 10 mg, 20mg
  Interventions: Drug: BF2.649
- Placebo (Placebo Comparator): Capsules of Placebo containing lactose with low, medium and high dosage
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BF2.649 — 1 capsule in the morning before breakfast
  Other Names: Pitolisant
  Arms: BF2.649
Drug: Placebo — 1 capsule in the morning before breakfast
  Arms: Placebo

SUMMARY:
Multicenter randomized double blind study versus placebo during 12 weeks with at first, an escalating dose period followed by stable dose period at the selected dose.

This double-blind period can be followed by a 9 months open-label period if the patient wishes to continue with the study product.

DETAILED DESCRIPTION:
The first period (12 weeks double blind period) will aim at demonstrating the efficacy and safety of BF2.649 by verifying whether the results of BF2.649 are superior to those of placebo.

The aim of the second period (open label extension phase) will be to assess the long-term tolerance, as well as the maintenance of the BF2.649 efficacy.

ELIGIBILITY:
Inclusion Criteria:

* patients with OSA treated by nCPAP but still complaining with EDS
* ESS score > or = 12

Exclusion Criteria:

* patient suffering from insomnia without OSA
* co-existing narcolepsy
* patient with sleep debt not due to OSA
* acute or chronic severe disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2011-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
ESS change (Epworth Sleepiness Scale) | at week 12 /52 versus baseline

CONTACTS AND LOCATIONS:
Overall Officials: Evelyne De Paillette, MD, Study Director — Bioprojet
Locations (1):
- CHU Grenoble, Grenoble, France

REFERENCES:
- [Derived] Pepin JL, Attali V, Causse C, Verbraecken J, Hedner J, Lecomte I, Tamisier R, Levy P, Lehert P, Dauvilliers Y. Long-Term Efficacy and Safety of Pitolisant for Residual Sleepiness Due to OSA. Chest. 2024 Mar;165(3):692-703. doi: 10.1016/j.chest.2023.11.017. Epub 2023 Nov 17. PMID 37979718
- [Derived] Pepin JL, Georgiev O, Tiholov R, Attali V, Verbraecken J, Buyse B, Partinen M, Fietze I, Belev G, Dokic D, Tamisier R, Levy P, Lecomte I, Lecomte JM, Schwartz JC, Dauvilliers Y; HAROSA I Study Group. Pitolisant for Residual Excessive Daytime Sleepiness in OSA Patients Adhering to CPAP: A Randomized Trial. Chest. 2021 Apr;159(4):1598-1609. doi: 10.1016/j.chest.2020.09.281. Epub 2020 Oct 26. PMID 33121980